CLINICAL TRIAL: NCT00897858
Title: Evaluation of Cerebral Spinal Fluid (CSF) Proteome and Angiogenesis Proteins in Children With Newly Diagnosed Central Nervous System Tumors
Brief Title: Studying Cerebrospinal Fluid Proteins and Angiogenesis Proteins in Young Patients With Newly Diagnosed Central Nervous System Tumors
Status: Withdrawn | Type: Observational
Why Stopped: This non-therapeutic study was registered in error. The PRS team doesn't delete studies once registered, so they recommended changing the status to Withdrawn
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000481330; PBTC-N08 (Other: Pediatric Brain Tumor Consortium)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; childhood atypical teratoid/rhabdoid tumor; untreated childhood visual pathway glioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; newly diagnosed childhood ependymoma; childhood craniopharyngioma; untreated childhood medulloblastoma; untreated childhood cerebellar astrocytoma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood brain stem glioma; untreated childhood visual pathway and hypothalamic glioma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Choroid Plexus Neoplasms; Rhabdoid Tumor; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric CNS tumor patients: Newly diagnosed pediatric patients with CNS tumor and no prior irradiation or chemotherapy

SUMMARY:
RATIONALE: Studying samples of cerebrospinal fluid from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer.

PURPOSE: This laboratory study is studying cerebrospinal fluid proteins and angiogenesis proteins in young patients with newly diagnosed central nervous system tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Investigate the feasibility of centrally collecting and processing high-quality cerebrospinal fluid (CSF) samples from pediatric patients with newly diagnosed central nervous system tumors for proteomic studies.
* Identify protein markers that might indicate the presence of a brain tumor using CSF samples collected from these patients.

OUTLINE: This is a multicenter study.

Patients undergo cerebrospinal fluid (CSF) collection from any or all of the following 5 sites: lumbar, cervical, ommaya, intra-operative (ventricular, cisternal), and/or external ventricular drain. CSF is obtained within 8 weeks of diagnosis but prior to (or concurrent with) the initiation of any post-operative therapy (excluding corticosteroids).

CSF samples are examined for proteomic biomarkers by 2D gel electrophoresis, low-mass fingerprinting, and stable isotope labeling.

PROJECTED ACCRUAL: A total of 99 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CNS tumors of any of the following histologies:

  * Diffuse pontine gliomas*
  * Focal/infiltrative tumors, including any of the following:

    * High- and low-grade gliomas
    * Gangliogliomas
    * Ependymomas
    * Oligodendrogliomas
    * Craniopharyngioma
    * Dysembryoplastic neuroepithelial tumors
    * Other low-grade neoplasms
  * Optic pathway gliomas*
  * Seeding tumors, including any of the following:

    * Germ cell tumors (germinomas and nongerminomas)
    * Embryonal tumors, including any of the following:

      * Medulloblastoma
      * Pineoblastoma
      * Supratentorial primitive neuroectodermal tumors
      * Atypical teratoid/rhabdoid tumor
      * Other embryonal tumors NOTE: *Histological requirement waived
* Newly diagnosed disease
* Cerebrospinal fluid (CSF) obtained as part of CSF diversion, initial diagnosis/staging, or administration of intrathecal chemotherapy (at the initiation of postoperative therapy)

PATIENT CHARACTERISTICS:

* Less than 22 years of age

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy
* Prior corticosteroids allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of newly diagnosed pediatric patients with a CNS tumor and no prior irradiation or chemotherapy. Cerebrospinal fluid (CSF) is withdrawn as part of initial diagnosis/staging, the administration of intrathecal therapy, or CSF diversion.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Number of IRB approvals of the study | Within 120 days of study release
  IRB approval will be used as a surrogate marker of support for this protocol.
Number of patients with proteomic data received at the Operations and Biostatistics Center | 12, 18, 24, and 30 months after 4th IRB approval
  Feasibility implies registering patients, submitting samples for proteomic investigation, and successfully analyzing the data at the lab in a timely fashion. The number of patients with proteomic data received at the PBTC Operations and Biostatistics Center will be assessed at 12, 18, 24, and 30 months after the 4th institution receives IRB approval for the study.
Number of differentially expressed biomarker proteins | Pre-treatment
  Unsupervised proteomic profiling will be done on the CSF samples obtained pre-treatment in order to identify proteins that differ between pediatric brain tumor patients and a banked set of pediatric control "normal" samples.

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Rood, MD, Study Chair — Children's National Research Institute
Locations (8):
- United States (8):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington